CLINICAL TRIAL: NCT05619809
Title: Chronic Thermogenic Dietary Supplement Consumption: Effects on Body Composition, Anthropometrics, Metabolism, and Subjective Variables
Brief Title: Chronic Thermogenic Dietary Supplement Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: EHP Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2022-933
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Body Composition Changes; Body Weight Changes; Anthropometric Changes; Metabolism Changes; Hemodynamic Changes
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermogenic Dietary Supplement (Experimental): Arm in which the thermogenic dietary supplement is consumed.
  Interventions: Dietary Supplement: Thermogenic dietary supplement; Dietary Supplement: Protein supplement
- Placebo Dietary Supplement (Placebo Comparator): Arm in which the placebo supplement is consumed.
  Interventions: Dietary Supplement: Protein supplement; Dietary Supplement: Placebo supplement
- Control (No Intervention): Control arm with no intervention.

INTERVENTIONS:
Dietary Supplement: Thermogenic dietary supplement — Daily ingestion of OxyShred thermogenic dietary supplement.
  Arms: Thermogenic Dietary Supplement
Dietary Supplement: Protein supplement — Daily ingestion of protein supplement.
  Arms: Placebo Dietary Supplement; Thermogenic Dietary Supplement
Dietary Supplement: Placebo supplement — Daily ingestion of a placebo dietary supplement.
  Arms: Placebo Dietary Supplement

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial. Healthy, exercising adult males and females will be recruited for participation. After providing informed consent, each participant will be randomized to one of three groups: 1) OxyShred thermogenic fat burner; 2) Placebo (PL); and 3) Control. All participants will complete a baseline laboratory visit consisting of assessments of body composition, anthropometry, metabolism, hemodynamics, dietary intake, exercise habits, and subjective variables. Participants in the two intervention groups (i.e., OxyShred and PL) will then be given dietary supplements for daily consumption, including OxyShred/PL and protein powder. Participants in all groups will complete the 4-week study and follow their usual training and nutrition habits - besides increased protein intake in the OxyShred and PL groups - along with questionnaires to assess compliance with the study protocol and potential side effects of supplementation. Following this 4-week period, participants will complete a second laboratory visit, where all baseline assessments will be repeated. The effects of group (OxyShred, PL, and control) and time (baseline, 4 weeks) will be statistically examined using linear models, along with appropriate post-hoc tests.

DETAILED DESCRIPTION:
Overview. This study is a randomized, double-blind, placebo-controlled trial. Healthy, exercising adult males and females will be recruited for participation. After providing informed consent, each participant will be randomized to one of three groups: 1) OxyShred thermogenic fat burner; 2) Placebo (PL); and 3) Control. All participants will complete a baseline laboratory visit consisting of assessments of body composition, anthropometry, metabolism, hemodynamics, dietary intake, exercise habits, and subjective variables. Participants in the two intervention groups (i.e., OxyShred and PL) will then be given dietary supplements for daily consumption, including OxyShred/PL and protein powder. Participants in all groups will complete the 4-week study and follow their usual training and nutrition habits - besides increased protein intake in the OxyShred and PL groups - along with questionnaires to assess compliance with the study protocol and potential side effects of supplementation. Following this 4-week period, participants will complete a second laboratory visit, where all baseline assessments will be repeated. The effects of group (OxyShred, PL, and control) and time (baseline, 4 weeks) will be statistically examined using linear models, along with appropriate post-hoc tests.

Participants. Eligible participants who provide consent will be stratified based on exercise training (resistance-trained, endurance-trained, or concurrently-trained), sex (male and female), and body composition (males: 10 to 20% vs. >20%; females: 15 to 25% vs. >25%), then randomly assigned to one of the three experimental groups (OxyShred, PL, or control) in a 2:2:1 ratio. Based on preliminary power analysis and comparison with previous studies, the target sample size is 50 participants (20 Oxyshred, 20 PL, and 10 control), with approximately equal representation of males and females.

Laboratory Visits. Participants will report to the laboratory at baseline and after 4 weeks of the assigned intervention. At both laboratory visits, participants will be interviewed to confirm adherence with pre-testing guidelines, such as fasting overnight and abstaining from food and fluid ingestion. Participants will then undergo body composition testing using the methods listed below. Anthropometric variables, such as waist circumference and wasit:hip ratio, will be collected via 3-dimensional optical scanning. Resting energy expenditure and substrate oxidation (respiratory quotient) will be assessed using indirect calorimetry, and resting heart rate and blood pressure will be quantified using an automated blood pressure monitor. Questionnaires will be used to assess physical activity levels, sleep, mood, and hunger related variables. The specific body composition assessment methods to be used are ADP (air displacement plethysmography), DXA (dual-energy x-ray absorptiometry), several bioelectrical impedance techniques, several 3-dimensional scanning techniques, ultrasound, and standard assessments of height and weight. All equipment will be calibrated as recommended by the device manufacturers each day prior to use. Metabolism will be assessed using indirect calorimetry. For the on-site surveys, the following questionnaires/surveys will be used: Demographics, Exercise Habits, and Caffeine Questionnaire; the International Physical Activity Questionnaire (IPAQ); the Pittsburgh Sleep Quality Index; the Mood and Feelings Questionnaire; the Three-Factor Eating Questionnaire (R18); ASA24; and menstrual cycle questionnaire for female participants. For the daily online compliance surveys, one of two forms will be used, depending on the group assignment of the participant.

Intervention. Participants randomized to the control group will be asked to continue their normal exercise and nutrition habits without making any modification for the duration of the study. However, as an incentive and to promote equity between conditions, control group participants will receive the protein supplement provided to the other groups after completion of the study. Participants in the OxyShred and PL group will be provided their assigned supplement (OxyShred or PL powder) along with supplemental protein, all provided by EHP labs. Oxyshred is a commercially available product, and the placebo will include the same flavoring agents and ingredients but without the active ingredients. The protein product is also commercially available. Participants will be asked to consume one dose of the OxyShred/PL supplement for the first week, either upon waking or 15 minutes prior to exercise, as indicated on product directions. After the first week, participants will be asked to consume two doses per day, one upon waking and one 15 minutes prior to exercise, which is also according to product directions. On days exercise is not performed, participants will be asked to consume one dose upon waking and a second dose in the early afternoon. Protein supplements will be provided to support body composition improvements. Participants with a baseline body mass between 50 and 59.9 kg will be asked to consume one serving (providing ~25 g protein) per day; participants with a baseline body mass between 60 and 89.9 kg will be asked to consume two servings per day (providing ~50 g protein); and participants with a baseline body mass between 90 and 110 kg will be asked to consume three servings per day (providing ~75 g protein). Besides the OxyShred/PL and protein supplementation, participants in the OxyShred and PL groups will be asked to generally continue their normal nutritional practices, including the types of foods they eat and eating frequency. However, all participants will be asked to refrain from consuming additional sports supplements and weight loss supplements throughout the trial. Consumption of general health support supplements, such as multivitamins, will be allowed if they were regularly consumed prior to study commencement (typically for ≥1 month). Daily caffeine intake, beyond that provided by the supplements, will be limited to ~100 mg per day, and participants will be provided with information about quantities of common foods or beverages providing this amount (e.g., one cup of coffee, two diet sodas, etc.). Throughout the intervention, compliance and potential side effects will be monitored via questionnaire. All participants will be asked to continue their typical exercise regimen and complete questionnaires documenting their frequency, duration, and type of exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 40
2. Non-smoker
3. Generally healthy based on self-report, defined as no known presence of uncontrolled disease or disorder, such as cardiovascular disease, metabolic disease, cancer, or musculoskeletal disorders; no major surgeries within the past 6 months; and no history of hypertension, coronary heart disease, angina, heart attack, stroke, or diabetes.
4. For those taking prescription medication, no changes in medication in the last month, nor any known limitations on consumption of caffeine or other supplements/substances contained in the dietary supplement alongside current medications.
5. Weight stable, defined as no changes in body weight greater than 4.5 kg in the past three months.
6. Exercise-trained, defined as performing exercise at least 2 times per week, on average, for the previous 6 months. Resistance-trained, endurance-trained, and concurrently-trained individuals will be eligible.
7. Moderate caffeine consumers, defined as an average daily intake of ~40 to 200 mg/d.
8. Body mass between 50 and 110 kg.
9. Body fat percentage ≥10% in males and ≥15% in females.
10. Willingness to comply with the experimental protocol, including consumption of dietary supplements and adherence to other study procedures.
11. Willingness to abstain from consumption from other sports supplements and weight loss supplements for the duration of the study.

Exclusion Criteria:

1. Failure to meet the aforementioned inclusion criteria
2. They self-report sensitivity to caffeine or other stimulants, including feelings of nervousness, jitteriness, and shakiness following consumption of doses of caffeine used in this study (i.e., 150 to 300 mg).
3. They are pregnant, currently trying to become pregnant, or breastfeeding.
4. They report allergy to any ingredient or component of any of the dietary supplements.
5. They self-report any other medical condition or consideration that the researchers believe could reasonably make participation unsafe, including the presence of a pacemaker or other electrical implant, claustrophobia, or other relevant conditions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Total body fat percentage | 4 weeks
  Total body fat percentage from dual-energy x-ray absorptiometry
Segmental body fat percentage | 4 weeks
  Segmental body fat percentage from dual-energy x-ray absorptiometry
Total fat mass | 4 weeks
  Total fat mass from dual-energy x-ray absorptiometry
Segmental fat mass | 4 weeks
  Segmental fat mass from dual-energy x-ray absorptiometry
Waist circumference | 4 weeks
  Waist circumference from 3-dimensional optical imaging
Waist-to-hip ratio | 4 weeks
  Waist-to-hip ratio from 3-dimensional optical imaging
Body mass | 4 weeks
  Body mass from scale

SECONDARY OUTCOMES:
Resting energy expenditure | 4 weeks
  Resting energy expenditure from indirect calorimetry
Respiratory quotient | 4 weeks
  Respiratory quotient from indirect calorimetry
Resting heart rate | 4 weeks
  Resting heart rate from automated sphygmomanometer
Resting blood pressure | 4 weeks
  Resting blood pressure from automated sphygmomanometer
Sleep quality | 4 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index
Mood ratings | 4 weeks
  Mood ratings as assessed by the Mood and Feelings Questionnaire
Eating behaviors | 4 weeks
  Eating behaviors as assessed by the Three-Factor Eating Questionnaire
Dietary intake | 4 weeks
  Dietary intake as assessed by the ASA24 recall method
Total lean soft tissue | 4 weeks
  Total lean soft tissue from dual-energy x-ray absorptiometry
Segmental lean soft tissue | 4 weeks
  Segmental lean soft tissue from dual-energy x-ray absorptiometry
Limb circumferences | 4 weeks
  Limb circumferences from 3-dimensional optical imaging
Side effects | 4 weeks
  Self-reported side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided